CLINICAL TRIAL: NCT01366521
Title: A Multicenter, Open-label, Dose Ranging Study to Determine the Pharmacokinetics and Pharmacodynamics of Mepolizumab Administered Intravenously or Subcutaneously to Adult Asthmatic Subjects With Elevated Blood Eosinophil Levels
Brief Title: Dose Ranging Pharmacokinetics and Pharmacodynamics Study With Mepolizumab in Asthma Patients With Elevated Eosinophils
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114092
Record Dates: First submitted 2011-05-12; First posted 2011-06-06 (Estimated); Results first posted 2015-12-10 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mepolizumab 250 mg subcutaneous (SC) (Experimental): 250 mg subcutaneous (SC)
  Interventions: Biological: Mepolizumab
- Mepolizumab 125 mg subcutaneous (SC) (Experimental): 125 mg subcutaneous (SC)
  Interventions: Biological: Mepolizumab
- Mepolizumab 12.5 mg subcutaneous (SC) (Experimental): 12.5 mg subcutaneous (SC)
  Interventions: Biological: Mepolizumab
- Mepolizimab 75 mg intravenously (I.V.) (Experimental): 75 mg intravenously (I.V.)
  Interventions: Biological: Mepolizumab

INTERVENTIONS:
Biological: Mepolizumab — Monoclonal antibody

SUMMARY:
A multi-center, randomized, open-label, parallel-group, repeat dose study in asthma patients with elevated eosinophils. Eligible subjects will receive 3 doses (28 days apart) of mepolizumab given intravenous (IV) or subcutaneously (SC). Blood samples for safety, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity analysis, as well as safety/tolerability assessments will be collected throughout the study

DETAILED DESCRIPTION:
Mepolizumab (SB-240563) is a humanized monoclonal antibody that blocks human interleukin 5 (IL-5) from binding to its receptor. Mepolizumab is currently under development for severe refractory asthma and a Phase IIB dose-ranging study using the IV route of administration is currently on-going. This study will be a multi-center, randomized, open-label, parallel-group, repeat dose study conducted in approximately 65 subjects with established asthma and elevated blood eosinophil levels. Dosing will occur on three occasions, every four weeks [Day 1, Day 28 (+/- 3 days) and Day 56 (+/- 3 days)]. Blood samples for safety, pharmacodynamics (PD), pharmacokinetics (PK) and immunogenicity analysis, as well safety and tolerability assessments will be collected/assessed throughout the study. Each subject will participate in the study for up to approximately 22 weeks, including screening, dosing and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Males or eligible females between 18 and 65 years of age inclusive, at the time of signing the informed consent; Non-childbearing potential is defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory]. To be eligible for entry into the study, females of child-bearing potential and females whose menopausal status is in question must commit to consistent and correct use of an acceptable method of birth control as defined in Section 7.1.1 from one month prior to the first dose of investigational product until 4 months after the last dose of investigational product.
* History of asthma for at least one year.
* Subjects must be on a stable dose of an inhaled corticosteroid or combination (ICS+LABA) therapy for at least 12 weeks prior to screening.
* FEV1≥45% and <90 % of predicted normal value during screening (obtained between 6:00 AM and 1:00 PM).
* Evidence of airway reversibility (FEV1≥12%) within 30 minutes of inhalation of albuterol OR airway hyperresponsiveness (PC20 of <8mg/mL or PD20 of <7.8 µ mol methacholine/histamine) documented in the 12 months prior to randomization.
* Subjects with documented evidence of elevated blood eosinophilia levels (>0.3 cells 109/L) within 12 months of screening and evidence of elevated blood eosinophilia levels (>0.3 cells 109/L) at screening.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* QTcF ≥450 msec; or QTcF ≥ 480 msec in subjects with Bundle Branch Block.
* AST, ALT, alkaline phosphatase and bilirubin ≥ 1.5xULN (isolated bilirubin <1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin ≥35%).
* Subjects with elevated blood eosinophil levels which is not related to asthma
* Current smokers (any subject who has smoked within the six months prior to screening or has a positive urine cotinine at screening) or subjects with a smoking history of >10 pack years calculated as follows:

Number of cigarettes per day X number of years smoked 20

* Presence of a clinically important lung condition other than asthma including current infection, bronchiectasis, pulmonary fibrosis, bronchopulmonary aspergillosis, Churg-Strauss syndrome, or diagnoses of emphysema or chronic bronchitis (chronic obstructive pulmonary disease other than asthma) or a history of lung cancer.
* An asthma exacerbation or respiratory tract infection within six weeks prior to screening (an exacerbation is defined as worsening asthma requiring the use of systemic corticosteroids and/or emergency department visit, hospitalisation).
* Subjects with a parasitic infestation within six months of screening.
* A current malignancy or previous history of cancer in remission for less than five years prior screening (except for localized carcinoma of the skin that has been resected for cure).
* Subjects who have clinically significant cardiovascular, endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, haematological or any other system abnormalities that are uncontrolled with standard treatment.
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices or persistent jaundice), cirrhosis, and known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Subjects with a known immunodeficiency (e.g. human immunodeficiency virus - HIV).
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within three months of screening.
* Subjects who have received omalizumab [Xolair] within 130 days of administration of the first dose of study medication.
* Subjects with recent history (within two years prior to screening) of alcohol misuse or substance abuse prior screening.
* A positive pre-study drug/alcohol test at screening.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, five half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Subjects who have previously participated in a study of mepolizumab and received study medication within 90 days prior to screening.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within seven days (or 14 days if the drug is a potential enzyme inducer) or five half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Exposure to live vaccine within the four weeks prior to screening and no intention to receive live vaccine during the study.
* History of sensitivity to the study medications (or components thereof) or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Pregnant or lactating females; pregnancy as determined by positive pregnancy test at screening or prior to dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (2):
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Pittsburgh, Pennsylvania
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (3):
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Pessac
- Germany (4):
  - GSK Investigational Site, Gauting, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114092 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114092 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114092 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114092 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114092 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114092 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114092 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) were on a stable dose of their current asthma medications for 12 weeks prior to screening. Par. who met the eligibility criteria at screening were randomized to one of the four possible treatment arms. Total duration of participation in the study was up to approximately 22 weeks including screening, dosing and follow-up.
Pre-assignment Details: A total of 70 participants were enrolled into the study and 66 participants completed the study.
Groups:
- Mepolizumab 12.5 mg SC: Participants received mepolizumab 12.5 milligrams (mg) administered subcutaneously (SC) (two injections of the same volume) once every 4 weeks (for a total of three doses on Day 1, Day 28 and Day 56). Maintenance asthma therapy was continued unchanged throughout the study, unless medically indicated.
- Mepolizumab 125 mg SC: Participants received mepolizumab 125 mg administered SC (two injections of the same volume) once every 4 weeks (for a total of three doses on Day 1, Day 28 and Day 56). Maintenance asthma therapy was continued unchanged throughout the study, unless medically indicated.
- Mepolizumab 250 mg SC: Participants received mepolizumab 250 mg administered SC (two injections of the same volume) once every 4 weeks (for a total of three doses on Day 1, Day 28 and Day 56). Maintenance asthma therapy was continued unchanged throughout the study, unless medically indicated.
- Mepolizumab 75 mg IV: Participants received mepolizumab 75 mg administered intravenously (IV) once every 4 weeks (for a total of three doses on Day 1, Day 28 and Day 56). Maintenance asthma therapy was continued unchanged throughout the study, unless medically indicated.
Period: Overall Study
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV
Started | 21 | 15 | 23 | 11
Completed | 20 | 14 | 21 | 11
Not Completed | 1 | 1 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV | Total
Number analyzed (Participants) | 21 | 15 | 23 | 11 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.1 (11.53) | 37.0 (17.80) | 43.9 (13.42) | 44.8 (12.55) | 42.3 (13.83)
Gender [Count of Participants; unit: Participants]
  Female | 13 | 5 | 14 | 5 | 37
  Male | 8 | 10 | 9 | 6 | 33
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1 | 0 | 1 | 0 | 2
  Asian-South East Asian Heritage | 0 | 1 | 1 | 0 | 2
  White-White/Caucasian/European Heritage | 20 | 14 | 21 | 11 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Blood Eosinophil Levels at Week 12 (Day 84)
Description: Change from Baseline in blood eosinophils was calculated as the post-Baseline value minus the Baseline value. The change from Baseline in log-transformed blood eosinophil levels at Week 12 was analyzed using both a linear and non-linear (Imax) dose response models. The dose response was found to be non-linear and hence only the results of the non-linear model are presented. Mepolizumab 75mg IV assumed to equate to 100 mg SC within model. Prior to log10-transformation, zero values were imputed with half the minimum value across all dose groups and time points. An adjustment for Baseline eosinophil count was also incorporated into the model.
Time Frame: Baseline (Day 1 pre-dose) and Week 12
Population: Pharmacodynamic (PD) Population: all participants randomized to treatment and who received at least one dose of study medication and who also had a Baseline PD or biomarker measurement and at least one post-treatment PD or biomarker measurement. Only participants who were available at the specified time point were analyzed.
Measure: Number (95% Confidence Interval); unit: Proportion of Baseline blood eosinophil
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV
Number analyzed (Participants) | 20 | 14 | 21 | 11
Proportion of Baseline blood eosinophil | 0.43 [0.31 to 0.58] | 0.14 [0.11 to 0.17] | 0.12 [0.10 to 0.15] | 0.14 [0.12 to 0.17]

2. Primary Outcome: Area Under the Blood Eosinophil Time Curve (AUEC) up to Day 84
Description: Area under the absolute blood eosinophil time curve to Day 84 (AUECeos[0-day 84]) determined using the linear trapezoidal rule for subset of participants with blood eosinophil data to Day 84. Blood samples for the analyses of AUEC(eos) (0-day 84) were collected at Days 1, 3, 7, 28, 56, 70 and 84.
Time Frame: Days 1, 3, 7, 28, 56, 70 and 84
Population: PD Population. Only participants with eosinophil data to Day 84 were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Giga unit per liter per day (GI*d/L)
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV
Number analyzed (Participants) | 20 | 14 | 21 | 11
Giga unit per liter per day (GI*d/L) | 21.551 [15.486 to 29.991] | 7.198 [5.290 to 9.796] | 6.381 [4.915 to 8.284] | 7.556 [5.459 to 10.459]

3. Primary Outcome: Maximum Change From Baseline in Blood Eosinophils (Emax)
Description: Blood samples were collected at Days 1, 3, 7, 28, 56, 70, 84, 112 and 140 to assess the maximum reduction from Baseline in blood eosinophils between Day 1 pre-dose and last quantifiable study measurement. Change from Baseline was calculated as the ratio of the post-Baseline value divided by the Baseline value. The maximum reduction from Baseline in eosinophils is represented by the minimum ratio to Baseline.
Time Frame: Days 1, 3, 7, 28, 56, 70, 84, 112 and 140
Population: PD Population
Measure: Geometric Mean (95% Confidence Interval); unit: Giga units per liter (GI/L)
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV
Number analyzed (Participants) | 21 | 15 | 23 | 11
Giga units per liter (GI/L) | 0.203 [0.124 to 0.331] | 0.113 [0.079 to 0.162] | 0.082 [0.057 to 0.119] | 0.141 [0.085 to 0.233]

4. Primary Outcome: Time to Maximum Change in Blood Eosinophils Levels (Tmaxeos)
Description: Blood samples were collected at Days 1, 3, 7, 28, 56, 70, 84, 112 and 140 to assess the time to first occurrence of maximum reduction from baseline in blood eosinophil levels between Day 1 pre-dose and last quantifiable study measurement.
Time Frame: Days 1, 3, 7, 28, 56, 70, 84, 112 and 140
Population: PD Population.
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV
Number analyzed (Participants) | 21 | 15 | 23 | 11
Days | 50.0 [34.6 to 65.5] | 49.4 [34.0 to 64.8] | 47.0 [32.0 to 62.0] | 58.8 [42.0 to 75.6]

5. Primary Outcome: Number of Participants Who Achieved >=50% Eosinophil Repletion by Day 140
Description: This summarizes the number of participants who returned to at least 50% of their Baseline blood eosinophil levels after maximum inhibition had been achieved and without any subsequent decrease in blood eosinophil levels. Blood samples were collected at Days 1, 3, 7, 28, 56, 70, 84, 112 and 140.
Time Frame: Days 1, 3, 7, 28, 56, 70, 84, 112 and 140
Population: PD Population
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV
Number analyzed (Participants) | 21 | 15 | 23 | 11
Participants | 8 | 1 | 2 | 1

6. Primary Outcome: Mean Area Under the Plasma-concentration Time Curve (AUC) Following SC and IV Administration of Mepolizumab
Description: AUC of mepolizumab was estimated by population modeling techniques using non-linear mixed effect methods for the individual and population pharmacokinetic parameters from the sparse sampling. Individual cumulative plasma of mepolizumab AUC to Day 84 (cumAUC(0-day 84)), is the sum of the AUCs over each dosing interval after each of the three doses administered, for those participants with data up to Day 84. Individual cumulative plasma of mepolizumab AUC to Day 140 (cumAUC(0-day 140) is the sum of the AUCs over each dosing interval after each of the three doses administered plus the AUC post the last dose interval up to Day 140 (i.e. from Day 84 to Day 140). Blood samples for PK analyses were collected on dosing days (Days 1, 28 and 56) at pre-dose and 0.5 hour (h), 1 h and 2 h post-dose (time was relative to the end of infusion in the IV cohort) as well as on Days 3, 7, 70, 84, 112 and 140 (follow-up visit).
Time Frame: Days 1, 3, 7, 28, 56, 70, 84, 112 and 140
Population: Pharmacokinetic (PK) Population: all participants randomized to treatment and who received at least one dose of study treatment and who have at least one PK sample taken and analyzed. Only those participants with the blood samples available at the indicated time points were analyzed (represented by n=X, X, X, X in the category titles).
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogramper milliliter per hour(ng*h/mL)
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV
Number analyzed (Participants) | 21 | 15 | 22 | 11
Nanogramper milliliter per hour(ng*h/mL)
  AUCtau, Dose1, n=21, 15, 22, 11 | 523632.6 [345804.8 to 792906.9] | 5091456.4 [4115689.6 to 6298562.4] | 8673608.7 [7635120.8 to 9853346.0] | 3986009.4 [3254498.2 to 4881941.8]
  AUCtau, Dose2, n=21, 14, 22, 11 | 793918.1 [516885.5 to 1219430.6] | 8391130.1 [7063697.1 to 9968018.6] | 13077585.6 [11596103.1 to 14748337.6] | 5959275.6 [4745685.2 to 7483211.5]
  AUCtau, Dose3, n=20, 14, 21, 11 | 908573.5 [586393.8 to 1407767.0] | 8837913.1 [7139982.5 to 10939621.6] | 14228122.9 [12457557.9 to 16250334.3] | 6714105.0 [5270701.1 to 8552791.3]

7. Primary Outcome: Maximum Plasma Concentration (Cmax) From Pre-dose (Day 1) to Day 140 for Mepolizumab
Description: Maximum plasma concentration was estimated by population modelling techniques using non-linear mixed effect methods for the individual and population pharmacokinetic parameters from the sparse sampling. Blood samples for PK analyses of mepolizumab were collected on dosing days (Days 1, 28 and 56) at pre-dose and 0.5 h, 1 h and 2 h post-dose (time was relative to the end of infusion in the IV cohort) as well as on Days 3, 7, 70, 84, 112 and 140 (follow-up visit).
Time Frame: Days 1, 3, 7, 28, 56, 70, 84, 112 and 140
Population: PK Population. Only those participants with the blood samples available at the indicated time points were analyzed (represented by n=X, X, X, X in the category titles).
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV
Number analyzed (Participants) | 21 | 15 | 22 | 11
Nanogram per milliliter (ng/mL)
  Cmax, Dose1, n=21, 15, 22, 11 | 1062.053 [672.280 to 1677.807] | 9904.234 [8108.129 to 12098.211] | 16112.461 [14138.105 to 18362.533] | 18103.887 [15189.165 to 21577.928]
  Cmax, Dose2, n=21, 14, 22, 11 | 1579.160 [1012.390 to 2463.228] | 14860.706 [12282.820 to 17979.633] | 24069.046 [21302.445 to 27194.952] | 21931.891 [18171.592 to 26470.320]
  Cmax, Dose3, n=20, 14, 21, 11 | 1784.626 [1134.380 to 2807.605] | 16574.716 [13650.258 to 20125.716] | 27307.211 [24043.561 to 31013.866] | 23576.215 [19424.780 to 28614.888]

8. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) From Pre-dose (Day 1) to Day 140 for Mepolizumab
Description: Time to maximum plasma concentration was estimated by population modelling techniques using non-linear mixed effect methods for the individual and population pharmacokinetic parameters from the sparse sampling. Blood samples for PK analyses of mepolizumab were collected on dosing days (Days 1, 28 and 56) at pre-dose and 0.5 h, 1 h and 2 h post-dose (time was relative to the end of infusion in the IV cohort) as well as on Days 3, 7, 70, 84, 112 and 140 (follow-up visit).
Time Frame: Days 1, 3, 7, 28, 56, 70, 84, 112 and 140
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV
Number analyzed (Participants) | 21 | 15 | 22 | 11
hours
  Tmax, Dose1, n=21, 15, 22, 11 | 200.490 [36.85 to 761.68] | 190.680 [105.82 to 457.17] | 193.665 [100.89 to 378.01] | 0.600 [0.50 to 0.75]
  Tmax, Dose2, n=21, 14, 22, 11 | 157.750 [37.50 to 503.39] | 148.780 [96.00 to 319.35] | 153.715 [87.29 to 263.83] | 0.500 [0.33 to 0.83]
  Tmax, Dose3, n=20, 14, 21, 11 | 143.310 [37.42 to 455.15] | 147.810 [93.42 to 256.29] | 140.940 [88.51 to 217.12] | 0.533 [0.42 to 0.75]

9. Primary Outcome: Terminal Half-life (t½) From Pre-dose (Day 1) to Day 140 for Mepolizumab
Description: Terminal half-life (t1/2) was estimated by modelling techniques using non-linear mixed effect methods for the individual and population pharmacokinetic parameters for mepolizumab from the sparse sampling. Blood samples for PK analyses of mepolizumab were collected on dosing days (Days 1, 28 and 56) at pre-dose and 0.5 h, 1 h and 2 h post-dose (time was relative to the end of infusion in the IV cohort) as well as on Days 3, 7, 70, 84, 112 and 140 (follow-up visit).
Time Frame: Days 1, 3, 7, 28, 56, 70, 84, 112 and 140
Population: PK Population
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV
Number analyzed (Participants) | 21 | 15 | 22 | 11
Days | 21.7676 [20.0070 to 23.5283] | 22.0979 [20.4834 to 23.7125] | 21.7561 [20.2230 to 23.2892] | 28.2336 [21.1455 to 35.3218]

10. Secondary Outcome: Number of Participants With Clinical Chemistry Parameters Outside the Normal Range Following Treatment
Description: Clinical chemistry laboratory parameters included blood urea nitrogen (BUN), potassium, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin (TB) and direct bilirubin, creatinine, chloride, uric acid, glucose, total carbondioxide (CO2), gamma glutamyltransferase (GGT), albumin, sodium, calcium, alkaline phosphatase (ALP) and total protein assessed at Baseline, Weeks 4, 8, 12 and 20. Laboratory abnormalities outside the normal range (high and low values) at any time post-Baseline are presented.
Time Frame: Baseline (Day 1 pre-dose), Weeks 4, 8, 12 and 20
Population: Safety Population: all participants randomized to treatment who received at least one dose of study medication. Only those participants available at the indicated time points were analyzed (represented by n=X, X, X, X in the category titles).
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV
Number analyzed (Participants) | 21 | 15 | 23 | 11
Participants
  Albumin, High, n=21,14,22,11 | 0 | 4 | 1 | 2
  ALP, High, n=21, 14, 22, 11 | 0 | 1 | 0 | 1
  ALP, Low, n=21, 14, 22, 11 | 1 | 0 | 0 | 0
  ALT, High, n=21, 14, 22, 11 | 1 | 0 | 2 | 3
  AST, High, n=21, 14, 22, 11 | 1 | 1 | 2 | 4
  TB, High, n=18, 14, 22, 11 | 0 | 1 | 0 | 0
  Calcium, High, n=21, 15, 23, 11 | 2 | 3 | 2 | 3
  Chloride, High, n=21, 14, 22, 11 | 6 | 5 | 6 | 3
  Chloride, Low, n=21, 14, 22, 11 | 0 | 0 | 0 | 1
  CO2 content/bicarbonate, Low, n=21, 14, 22, 11 | 8 | 4 | 7 | 6
  Creatinine, High, n=21, 14, 22, 11 | 1 | 0 | 0 | 0
  Creatinine, Low, n=21, 14, 22, 11 | 4 | 2 | 5 | 2
  GGT, High, n=21, 14, 22, 11 | 3 | 0 | 3 | 6
  Glucose, High, n=21, 15, 23, 11 | 5 | 7 | 5 | 5
  Glucose, Low, n=21, 15, 23, 11 | 1 | 2 | 5 | 1
  Potassium, Low, n=20, 14, 21, 11 | 0 | 1 | 0 | 1
  Sodium, High, n=20, 14, 21, 11 | 0 | 0 | 1 | 0
  Sodium, Low, n=20, 14, 21, 11 | 0 | 0 | 1 | 1
  Total Protein, High, n=18, 14, 21, 10 | 0 | 0 | 0 | 1
  Urea/BUN, High, n=20, 14, 21, 11 | 2 | 1 | 1 | 0
  Urea/BUN, Low, n=20, 14, 21, 11 | 0 | 0 | 1 | 0
  Uric acid, High, n=21, 14, 22, 11 | 1 | 2 | 0 | 3
  Uric acid, Low, n=21, 14, 22, 11 | 0 | 0 | 0 | 1

11. Secondary Outcome: Number of Participants With Hematology Laboratory Parameters Outside the Normal Range at Following Treatment
Description: Hematology laboratory parameters included platelet count, red blood cells (RBC) count, white blood cell (WBC) count, hemoglobin, hematocrit, reticulocyte count, mean corpuscle volume (MCV), mean corpuscle hemoglobin (MCH), mean corpuscle hemoglobin concentration (MCHC), neutrophils, segmented neutrophils (SN), total neutrophils (TN), lymphocytes, monocytes, eosinophils and basophils assessed at Baseline, Weeks 4, 8, 12 and 20. Hematology abnormalities outside the normal range (high and low values) at any time post-Baseline are presented.
Time Frame: Days 1, 3, 7, 28, 56, 70, 84, 112 and 140 (follow-up visit)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV
Number analyzed (Participants) | 21 | 15 | 23 | 11
Participants
  Eosinophils, High | 10 | 2 | 2 | 0
  Eosinophils, Low | 4 | 6 | 11 | 4
  Eosinophils percentage, High | 12 | 1 | 3 | 0
  Hemoglobin, High | 1 | 0 | 1 | 2
  Hemoglobin, Low | 5 | 3 | 2 | 2
  Hematocrit, High | 2 | 0 | 1 | 1
  Hematocrit, Low | 5 | 2 | 2 | 2
  Lymphocytes, High | 0 | 0 | 0 | 1
  Lymphocytes, Low | 2 | 0 | 3 | 1
  Lymphocytes-percentage, High | 4 | 5 | 2 | 3
  Lymphocytes-percentage, Low | 2 | 0 | 7 | 3
  MCHC, Low | 6 | 2 | 4 | 0
  MCH, High | 3 | 3 | 2 | 3
  MCH, Low | 2 | 0 | 1 | 0
  MCV, High | 2 | 3 | 0 | 2
  Monocytes, High | 0 | 1 | 0 | 0
  Monocytes, Low | 7 | 2 | 3 | 2
  Monocytes percentage, High | 3 | 3 | 3 | 0
  SN, High | 3 | 0 | 3 | 2
  SN, Low | 4 | 4 | 4 | 1
  SN-percentage, High | 6 | 2 | 8 | 3
  SN-percentage, Low | 5 | 4 | 1 | 1
  TN, High | 3 | 0 | 3 | 2
  TN, Low | 4 | 4 | 4 | 1
  TN-percentage, High | 6 | 2 | 8 | 3
  TN-percentage, Low | 5 | 4 | 1 | 1
  Platelet count, High | 0 | 1 | 2 | 0
  Platelet count, Low | 0 | 1 | 1 | 0
  RBC, High | 0 | 0 | 1 | 1
  RBC, Low | 6 | 4 | 2 | 3
  Reticulocytes count, High | 4 | 2 | 9 | 8
  Reticulocytes count, Low | 10 | 3 | 8 | 0
  WBC, High | 5 | 1 | 1 | 3
  WBC, Low | 2 | 4 | 3 | 1

12. Secondary Outcome: Change From Baseline in Systolic Blood Pressure and Diastolic Blood Pressure Assessed at Baseline, Day 1, Day 28, Day 56, Day 84, Day 112 and Day 140
Description: Vital sign measurements including systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured at Baseline (pre-dose Day 1), Day 1 (30 minutes, 1 h, 2 h), Day 28 (pre-dose, 30 minutes, 1 h, 2 h), Day 56 (pre-dose, 30 minutes, 1 h, 2 h), Day 84, Day 112 and follow-up (Day 140).
Time Frame: Baseline (Day 1 pre-dose) and at Day 1, Day 28, Day 56, Day 84, Day 112 and Day 140
Population: Safety Population. Only those participants available at the indicated time points were analyzed (represented by n=X, X, X, X in the category titles).
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV
Number analyzed (Participants) | 21 | 15 | 23 | 11
Millimeter of mercury (mmHg)
  SBP, Day 1, 30 min, n=21,15,23,11 | 0.0 (8.30) | -4.0 (13.32) | 1.0 (6.91) | 0.3 (5.64)
  SBP, Day 1,1 H, n=21,15,23,11 | 0.1 (9.26) | -2.9 (13.26) | 1.3 (9.46) | 0.0 (7.80)
  SBP, Day 1, 2 H, n=21,15,23,11 | 0.2 (10.26) | 0.2 (14.31) | 2.0 (8.69) | 0.0 (8.19)
  SBP, Day 28, pre-dose, n=21,14,22,11 | -2.5 (11.46) | -7.6 (9.50) | -0.8 (10.24) | 4.0 (11.58)
  SBP, Day 28, 30 min, n=21,14,22,11 | 1.9 (13.39) | -9.0 (9.12) | -0.3 (11.44) | 1.6 (12.59)
  SBP, Day 28, 1 H, n=21,14,22,11 | -0.7 (12.67) | -9.8 (10.81) | -0.3 (11.00) | 1.9 (10.72)
  SBP, Day 28, 2 H, n=21,14,22,11 | 2.8 (12.89) | -6.3 (12.22) | 0.7 (8.89) | 4.7 (9.82)
  SBP, Day 56, pre-dose, n=20,14,21,11 | -2.0 (11.50) | -3.7 (11.26) | -1.0 (12.09) | 1.0 (10.17)
  SBP, Day 56, 30 min, n=20,14,21,11 | -1.8 (11.93) | -5.0 (13.11) | 0.3 (10.47) | 1.8 (9.31)
  SBP, Day 56, 1 H, n=20,14,21,11 | -3.7 (12.58) | -3.5 (12.38) | -0.2 (15.04) | -0.4 (8.29)
  SBP, Day 56, 2 H, n=20,14,21,11 | 0.1 (12.76) | -5.0 (14.38) | 3.7 (13.54) | 3.5 (9.17)
  SBP, Day 84, n=20,14,21,11 | 1.6 (12.42) | -7.9 (11.73) | 0.0 (10.61) | 0.5 (8.48)
  SBP, Day 112, n=20,14,21,11 | 0.4 (11.32) | -1.6 (12.77) | -1.4 (11.02) | 0.8 (12.80)
  SBP, Follow-up, n=20,14,21,11 | 2.2 (14.33) | -0.9 (15.13) | -1.0 (12.52) | 3.3 (9.45)
  DBP, Day 1, 30 min, n=21,15,23,11 | -1.1 (5.22) | -2.1 (11.63) | -0.9 (7.29) | -0.9 (6.70)
  DBP, Day 1,1 H, n=21,15,23,11 | -2.0 (5.77) | -3.3 (11.12) | -2.1 (7.46) | -3.7 (4.31)
  DBP, Day 1, 2 H, n=21,15,23,11 | -0.7 (5.26) | 0.1 (10.27) | 0.3 (8.36) | -1.6 (6.77)
  DBP, Day 28, pre-dose, n=21,14,22,11 | -1.4 (9.21) | -3.6 (8.22) | -1.8 (9.17) | -3.7 (14.07)
  DBP, Day 28, 30 min, n=21,14,22,11 | -0.7 (9.25) | -3.4 (8.43) | 0.0 (12.15) | -3.6 (12.92)
  DBP, Day 28, 1 H, n=21,14,22,11 | -4.0 (8.95) | -4.4 (10.43) | -3.2 (9.78) | -3.5 (12.91)
  DBP, Day 28, 2 H, n=21,14,22,11 | 1.1 (8.35) | -3.9 (10.36) | -0.7 (9.73) | -3.9 (13.95)
  DBP, Day 56, pre-dose, n=20,14,21,11 | 0.8 (6.24) | -0.1 (8.19) | -3.2 (7.57) | -1.9 (11.47)
  DBP, Day 56, 30 min, n=20,14,21,11 | -0.4 (8.32) | -0.9 (11.18) | -1.8 (7.03) | -1.9 (12.19)
  DBP, Day 56, 1 H, n=20,14,21,11 | -0.8 (7.37) | -0.8 (10.87) | -3.7 (6.34) | -4.0 (11.37)
  DBP, Day 56, 2 H, n=20,14,21,11 | 2.1 (8.26) | -0.4 (11.24) | 0.1 (9.65) | -2.1 (10.30)
  DBP, Day 84, n=20,14,21,11 | -0.6 (8.56) | -2.4 (8.79) | -1.7 (7.90) | -1.4 (10.94)
  DBP, Day 112, n=20,14,21,11 | 0.3 (8.07) | 1.9 (13.20) | -2.8 (10.65) | 0.8 (13.59)
  DBP, Follow-up, n=20,14,21,11 | 1.3 (8.63) | 4.0 (10.86) | -1.6 (11.38) | -2.3 (9.74)

13. Secondary Outcome: Change From Baseline in Heart Rate Assessed at Baseline, Day 1, Day 28, Day 56, Day 84, Day 112 and Day 140
Description: Vital sign measurements including heart rate (HR) was measured at Baseline (Pre-dose Day 1), Day 1 (30 minutes, 1 h, 2 h), Day 28 (pre-dose, 30 minutes, 1 h, 2 h), Day 56 (pre-dose, 30 minutes, 1 h, 2 h), Day 84, Day 112 and follow-up (Day 140).
Time Frame: Baseline (Day 1 pre-dose) and at Day 1, Day 28, Day 56, Day 84, Day 112 and Day 140
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: beats per minute (BPM)
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV
Number analyzed (Participants) | 21 | 15 | 23 | 11
beats per minute (BPM)
  HR, Day 1, 30 min, n=21,15,23,11 | -2.7 (5.35) | -3.7 (9.37) | -2.1 (7.51) | 1.1 (7.08)
  HR, Day 1,1 H, n=21,15,23,11 | -3.2 (6.69) | -3.9 (9.88) | -1.9 (7.00) | 1.9 (5.89)
  HR, Day 1, 2 H, n=21,15,23,11 | -1.7 (7.36) | -3.3 (7.22) | -0.4 (6.21) | 11.3 (21.47)
  HR, Day 28, pre-dose, n=21,14,22,11 | 1.6 (10.82) | -2.5 (11.27) | -0.1 (9.80) | 1.1 (8.38)
  HR, Day 28, 30 min, n=21,14,22,11 | 1.8 (7.83) | -3.4 (11.21) | -2.2 (10.35) | 3.2 (11.96)
  HR, Day 28, 1 H, n=21,14,22,11 | 1.3 (10.22) | -4.2 (10.53) | -2.0 (11.54) | 1.9 (11.48)
  HR, Day 28, 2 H, n=21,14,22,11 | 0.1 (7.70) | -2.2 (9.93) | 1.4 (10.60) | 2.5 (12.07)
  HR, Day 56, pre-dose, n=20,14,21,11 | 3.8 (11.41) | -3.3 (10.32) | -0.4 (10.13) | 2.5 (8.12)
  HR, Day 56, 30 min, n=20,14,21,11 | 0.3 (10.08) | -3.3 (11.84) | -1.0 (10.85) | -0.4 (9.29)
  HR, Day 56, 1 H, n=20,14,21,11 | 0.5 (9.71) | -3.4 (12.64) | 0.3 (11.01) | 2.0 (8.49)
  HR, Day 56, 2 H, n=20,14,21,11 | 1.7 (10.15) | -4.1 (15.73) | -0.1 (9.83) | 4.5 (15.21)
  HR, Day 84, n=20,14,21,11 | 1.9 (9.37) | -0.1 (8.10) | 2.6 (10.53) | 4.3 (12.11)
  HR, Day 112, n=20,14,21,11 | 2.7 (10.72) | -3.3 (12.48) | 2.4 (11.97) | 2.5 (8.10)
  HR, Follow-up, n=20,14,21,11 | 2.4 (10.29) | -1.7 (10.77) | 1.1 (8.78) | 7.0 (15.13)

14. Secondary Outcome: Number of Participants With Levels of Anti-mepolizumab Antibodies at Indicated Time Points
Description: Blood samples were collected for the determination of anti-mepolizumab antibodies by antibody detection (AD) and antibody neutralisation (AN) assay. For participants who prematurely withdrew from the study and had been dosed, immunogenicity testing occurred (if possible) at the time of premature withdrawal and at 16 weeks after dosing (or the end of the study, whichever came first). Serum was tested for the presence of anti-mepolizumab antibodies using the currently approved analytical methodology incorporating screening, confirmation and titration steps. Samples confirmed positive for the presence of anti-mepolizumab antibodies in the original assay were tested for the presence of neutralizing antibodies.
Time Frame: Day 1, Day 112 and Day 140
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV
Number analyzed (Participants) | 21 | 15 | 23 | 11
Participants
  Day 1, AD-positive, n=21,15,22,11 | 1 | 1 | 0 | 0
  Day 1, AN-Negative, n=1,1,0,0 | 1 | 1 | 0 | 0
  Day 112, AD-Positive, n=20,13,21,11 | 1 | 2 | 3 | 0
  Day 112, AN-Negative, n=1,2,3,0 | 1 | 2 | 3 | 0
  Follow-up, AD-Positive, n=20,14,21,10 | 2 | 1 | 2 | 0
  Follow-up, AN-Negative, n=2,1,2,0 | 2 | 1 | 2 | 0

15. Secondary Outcome: Number of Participants With the Indicated Electrocardiogram (ECG) Findings at Screening and Day 3
Description: The number of participants with normal, abnormal - clinically significant (CS), and abnormal - not clinically significant (NCS) ECG findings, as well as the number of participants with no results (NR), at Screening (SCR) and Day 3 are presented. Findings were determined to be normal, abnormal CS, and NCS by the investigator.
Time Frame: Screening (SCR) and at Day 3
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab 75 mg IV
Number analyzed (Participants) | 21 | 15 | 23 | 11
Participants
  SCR, Normal, n=21, 15, 23, 11 | 17 | 12 | 19 | 6
  SCR, NCS, n=21, 15, 23, 11 | 4 | 2 | 4 | 5
  SCR, NR, n=21, 15, 23, 11 | 0 | 1 | 0 | 0
  Day 3, Normal, n=20, 14, 22, 11 | 15 | 11 | 16 | 7
  Day 3, NCS, n=20, 14, 22, 11 | 5 | 3 | 6 | 4

16. Secondary Outcome: Mean AUC to Assess the Absolute Bioavailability of SC Mepolizumab
Description: Population modelling techniques using non-linear mixed effect methods were used to estimate individual and population pharmacokinetic parameters from the sparse sampling. Log-transformed individual clearance estimates were analysed using an analysis of variance (ANOVA) model. The absolute bioavailability for each SC dose group and across SC doses will be estimated from the model together with associated 90% confidence intervals. Blood samples for PK analyses were collected on dosing days (Days 1, 28 and 56) at pre-dose and 0.5 h, 1 h and 2 h post-dose (time was relative to the end of infusion in the IV cohort) as well as on Days 3, 7, 70, 84, 112 and 140 (follow-up visit).
Time Frame: Days 1, 3, 7, 28, 56, 70, 84, 112 and 140
Population: PK Population
Measure: Mean (90% Confidence Interval); unit: Percentage
Groups:
- Mepolizumab SC Overall: Combined results for participants receiving either mepolizumab 12.5 mg, 125 mg or 250 mg administered SC (two injections of the same volume) once every 4 weeks (for a total of three doses on Day 1, Day 28 and Day 56). Maintenance asthma therapy was continued unchanged throughout the study, unless medically indicated.
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab SC Overall
Number analyzed (Participants) | 21 | 15 | 22 | 58
Percentage | 81.04 [56.50 to 116.23] | 81.59 [55.54 to 119.85] | 63.82 [44.62 to 91.28] | 74.15 [53.92 to 101.97]

17. Secondary Outcome: Mean Dose Normalized Cmax Ratio to Assess the Relative Bioavailability of SC Mepolizumab as Compared With IV Mepolizumab
Description: Maximum plasma concentration was estimated by population modelling techniques using non-linear mixed effect methods for the individual and population pharmacokinetic parameters from the sparse sampling. Log-transformed dose-normalized (DM) Cmax were be analyzed using an analysis of variance (ANOVA) model. The ratio for each SC dose group versus IV and across SC doses versus IV will be estimated from the model together with associated 90% confidence intervals. Blood samples for PK analyses of mepolizumab were collected on dosing days (Days 1, 28 and 56) at pre-dose and 0.5 h, 1 h and 2 h post-dose (time was relative to the end of infusion in the IV cohort) as well as on Days 3, 7, 70, 84, 112 and 140 (follow-up visit).
Time Frame: Days 1, 3, 7, 28, 56, 70, 84, 112 and 140
Population: PK Population. Only those participants available at the indicated time points were analyzed (represented by n=X, X, X, X in the category titles).
Measure: Mean (90% Confidence Interval); unit: Percentage
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab SC Overall
Number analyzed (Participants) | 21 | 15 | 22 | 58
Percentage
  DM Cmax ratio (first dose), n=21, 15, 22, 58 | 46.93 [32.05 to 68.73] | 43.77 [29.14 to 65.74] | 35.60 [24.38 to 51.98] | 41.50 [29.63 to 58.14]
  DM Cmax ratio (third dose), n=20, 14, 21, 55 | 60.56 [41.80 to 87.72] | 56.24 [37.78 to 83.72] | 46.33 [32.08 to 66.90] | 53.65 [38.72 to 74.34]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and Serious adverse events (SAEs) were collected from the administration of the first dose of study medication and until the final follow-up contact (up to Week 20).
Description: AEs and SAEs were collected in participants of the Safety Population, comprised of all participants randomized to treatment who received at least one dose of study medication.
Arm/Group | Mepolizumab 12.5 mg SC | Mepolizumab 125 mg SC | Mepolizumab 250 mg SC | Mepolizumab SC Overall | Mepolizumab 75 mg IV
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/15 | 0/23 | 1/59 | 0/11
Other Adverse Events (participants affected / at risk) | 14/21 | 7/15 | 12/23 | 33/59 | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mepolizumab 12.5 mg SC (N=21) | Mepolizumab 125 mg SC (N=15) | Mepolizumab 250 mg SC (N=23) | Mepolizumab SC Overall (N=59) | Mepolizumab 75 mg IV (N=11)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mepolizumab 12.5 mg SC (N=21) | Mepolizumab 125 mg SC (N=15) | Mepolizumab 250 mg SC (N=23) | Mepolizumab SC Overall (N=59) | Mepolizumab 75 mg IV (N=11)
Nasopharyngitis (Infections and infestations) | 3 | 1 | 2 | 6 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 3 | 3 | 1 | 7 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 2 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 1 | 0
Irritability (General disorders) | 1 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 6 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Burn oesophageal (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 2 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Heart rate increased (Investigations) | 0 | 1 | 0 | 1 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.